CLINICAL TRIAL: NCT07108530
Title: Integrated Treatment Protocol for Induction/Consolidation Chemotherapy and Transplantation in Adult Acute Myeloid Leukemia Multicenter Study on the Efficacy of an Integrated Treatment Approach
Brief Title: Efficacy of Integrated Induction-Consolidation Chemotherapy and Transplantation for Adult Acute Myeloid Leukemia: Multicenter Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanxiBethuneH2
Record Dates: First submitted 2025-07-01; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — DAV regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficacy of Integrated Induction-Consolidation Chemotherapy and Transplantation for Adult Acute Myel (Experimental)
  Interventions: Other: Integrated IAV/MA Chemotherapy and Allo-HSCT Protocol for Adult AML; Drug: First Induction (IAV or DAV Regimen); Drug: Consolidation Therapy Options: MA or Intermediate-Dose Cytarabine Regimen; Other: Subsequent Treatment Plan for Transplant-Eligible Patients; Other: Allogeneic Stem Cell Transplantation Protocol; Other: GVHD Prophylaxis Regimen; Other: Subsequent Consolidation Therapy for Transplant-Ineligible Patients

INTERVENTIONS:
Other: Integrated IAV/MA Chemotherapy and Allo-HSCT Protocol for Adult AML — This intervention is distinguished by its risk-adapted, time-compressed, and economically tiered design. It integrates two induction options-IAV (idarubicin + cytarabine + venetoclax) for patients with better economic resources and DAV (daunorubicin + cytarabine + venetoclax) for those with limited resources-followed by consolidation with either the MA regimen (liposomal mitoxantrone + intermediate-dose cytarabine) or intermediate-dose cytarabine alone. Eligible patients proceed directly to allogeneic hematopoietic stem cell transplantation (allo-HSCT) with a FA-BuCy/ATG conditioning regimen and a novel GVHD prophylaxis strategy using anti-CD25 monoclonal antibody combined with delayed oral cyclosporine. The entire treatment is designed to be completed within four months from diagnosis. This protocol is unique in its combination of liposomal chemotherapy, venetoclax-based induction, and tailored transplant strategies.
Drug: First Induction (IAV or DAV Regimen) — * IAV Regimen:Intravenous Idarubicin (Ida): 6 mg/m²/day on days 1-3 (total cumulative dose ≤ 40 mg)，Intravenous Cytarabine: 100 mg/m²/day on days 1-7，Oral Venetoclax: 8-day schedule（100 mg on day 4, 200 mg on day 5, and 400 mg/day on days 6-11）
  * DAV Regimen：Intravenous Daunorubicin (D): 60 mg/m²/day on days 1-3，Intravenous Cytarabine: 100 mg/m²/day on days 1-7，Oral Venetoclax: 8-day schedule（100 mg on day 4, 200 mg on day 5, and 400 mg/day on days 6-11）
Drug: Consolidation Therapy Options: MA or Intermediate-Dose Cytarabine Regimen — * MA Regimen (Liposomal Mitoxantrone + Intermediate-Dose Cytarabine):Liposomal Mitoxantrone: 10 mg/m²/day on days 1-2.Cytarabine: 1 g/m² every 12 hours for 3 days (days 1-3).
  * Intermediate-Dose Cytarabine Regimen:Cytarabine: 1 g/m² every 12 hours for 3 days (days 1-3).
Other: Subsequent Treatment Plan for Transplant-Eligible Patients — Patients eligible for allogeneic hematopoietic stem cell transplantation (allo-HSCT) should proceed directly to transplant after the above two treatment cycles（The requirement before transplantation is that minimal residual disease should be negative).
  * Conditioning Regimen: FA + BuCy (Fludarabine + Busulfan + Cyclophosphamide). For haploidentical transplantation, ATG (antithymocyte globulin) is added.
  * Donor Selection Priority:
    1. HLA-matched sibling donor (MSD)
    2. Matched unrelated donor (MUD)
    3. Haploidentical donor (Haplo) Selection should consider donor age, health status, and other clinical factors.
Other: Allogeneic Stem Cell Transplantation Protocol — Conditioning Regimen: FA-BuCy/ATG
  * Fludarabine: 30 mg/m²/day on days -8 to -6
  * Cytarabine: 1 g/m²/day on days -8 to -6
  * Busulfan: 2.4 mg/kg/day on days -5 to -3
  * Cyclophosphamide: 30 mg/kg/day on days -4 to -3
  * ATG (Antithymocyte Globulin): 7.5 mg/kg total dose, administered from day -5 to -2
Other: GVHD Prophylaxis Regimen — GVHD Prophylaxis
  * Recombinant Humanized Anti-CD25 Monoclonal Antibody: 50 mg on days +1 and +4.
  * The GVHD prophylaxis regimen consists of cyclosporine, mycophenolate mofetil (MMF), and short-course methotrexate (MTX).Cyclosporine (CsA):Initiated as a continuous 24-hour intravenous infusion at a dose of 2 mg/kg/day, starting from day -9 before transplantation.Once the patient can tolerate oral intake, cyclosporine is switched to oral administration at a dose of 3-5 mg/kg/day, divided into two daily doses.The target therapeutic trough concentration of cyclosporine should be maintained between 150-250 μg/L.
  * Delayed Oral Cyclosporine Protocol:Continue IV infusion until day +20, even if GI symptoms resolve.Switch to oral only if no acute GVHD occurs.If grade II-IV acute GVHD develops, continue IV CsA.
Other: Subsequent Consolidation Therapy for Transplant-Ineligible Patients — 1. Consolidation Therapy (Two Cycles)
     * Option A Intermediate-Dose Cytarabine-Based Regimen：Liposomal Mitoxantrone: 10 mg/day on days 1-2 (dose-reduced).Cytarabine: 1 g/m² every 12 hours for 3 days (days 1-3).
     * Option B VA Regimen (Venetoclax + Azacitidine)：Venetoclax (V): Dose-escalation starting at 100 mg on day 1, increasing to 400 mg/day by day 6, continued through day 14.Azacitidine (A): 75 mg/m²/day subcutaneously or intravenously on days 1-7.
     * Treatment Cycle:Each regimen is administered for two cycles with a 3-week interval between cycles, followed by maintenance therapy.
  2. Maintenance Therapy After Two Consolidation Cycles
     * Pegylated Interferon α-2b (Long-acting Interferon): 180μg subcutaneously every two weeks.
  Continued until disease progression or unacceptable toxicity occurs.

SUMMARY:
This is a multicenter, single-arm, open-label clinical study designed to evaluate the efficacy and safety of an integrated "induction-consolidation-transplantation" treatment protocol in adult patients with acute myeloid leukemia (AML, excluding M3 subtype). Based on patients' economic conditions, two induction regimens are offered: the IAV regimen (idarubicin + cytarabine + venetoclax) for those with better financial resources, and the DAV regimen (daunorubicin + cytarabine + venetoclax) for those with limited resources. During the consolidation phase, patients receive either the MA regimen (liposomal mitoxantrone + intermediate-dose cytarabine) or intermediate-dose cytarabine monotherapy. Eligible patients proceed directly to allogeneic hematopoietic stem cell transplantation (allo-HSCT), with a FA-BuCy/ATG conditioning regimen and an innovative graft-versus-host disease (GVHD) prophylaxis strategy using anti-CD25 monoclonal antibody combined with delayed oral cyclosporine. The entire treatment plan is designed to be completed within four months of diagnosis. The study plans to enroll 50 newly diagnosed patients aged 14-65 years. Primary endpoints include disease-free survival (DFS), complete remission rate (CR/CRi), and the efficacy of the transplantation protocol. Secondary endpoints include relapse rate, treatment-related mortality, 2-year overall survival, and treatment safety. This study aims to explore a new strategy to improve the cure rate of AML by optimizing drug combinations and shortening the treatment duration.

DETAILED DESCRIPTION:
Intervention Measures

1. Induction and Consolidation Treatment Regimen 1.1 First Induction Therapy: IAV or DAV Regimen

   * IAV Regimen:Intravenous Idarubicin (Ida): 6 mg/m²/day on days 1-3 (total cumulative dose ≤ 40 mg)，Intravenous Cytarabine: 100 mg/m²/day on days 1-7，Oral Venetoclax: 8-day schedule（100 mg on day 4, 200 mg on day 5, and 400 mg/day on days 6-11）
   * DAV Regimen：Intravenous Daunorubicin (D): 60 mg/m²/day on days 1-3，Intravenous Cytarabine: 100 mg/m²/day on days 1-7，Oral Venetoclax: 8-day schedule（100 mg on day 4, 200 mg on day 5, and 400 mg/day on days 6-11） 1.2 Consolidation Therapy Options: MA or Intermediate-Dose Cytarabine Regimen
   * MA Regimen (Liposomal Mitoxantrone + Intermediate-Dose Cytarabine):Liposomal Mitoxantrone: 10 mg/m²/day on days 1-2.Cytarabine: 1 g/m² every 12 hours for 3 days (days 1-3).
   * Intermediate-Dose Cytarabine Regimen:Cytarabine: 1 g/m² every 12 hours for 3 days (days 1-3).

   Summary:
   * For patients with good economic conditions: IAV → MA regimen.
   * For patients with limited economic resources: DAV → Intermediate-dose cytarabine regimen.
2. Subsequent Treatment Plan for Transplant-Eligible Patients Patients eligible for allogeneic hematopoietic stem cell transplantation (allo-HSCT) should proceed directly to transplant after the above two treatment cycles（The requirement before transplantation is that minimal residual disease should be negative).

   * Conditioning Regimen: FA + BuCy (Fludarabine + Busulfan + Cyclophosphamide). For haploidentical transplantation, ATG (antithymocyte globulin) is added.
   * Donor Selection Priority:

1. HLA-matched sibling donor (MSD) 2. Matched unrelated donor (MUD) 3. Haploidentical donor (Haplo) Selection should consider donor age, health status, and other clinical factors. 3.Allogeneic Stem Cell Transplantation Protocol 3.1 Conditioning Regimen: FA-BuCy/ATG

* Fludarabine: 30 mg/m²/day on days -8 to -6
* Cytarabine: 1 g/m²/day on days -8 to -6
* Busulfan: 2.4 mg/kg/day on days -5 to -3
* Cyclophosphamide: 30 mg/kg/day on days -4 to -3
* ATG (Antithymocyte Globulin): 7.5 mg/kg total dose, administered from day -5 to -2 3.2 GVHD Prophylaxis
* Recombinant Humanized Anti-CD25 Monoclonal Antibody: 50 mg on days +1 and +4.
* The GVHD prophylaxis regimen consists of cyclosporine, mycophenolate mofetil (MMF), and short-course methotrexate (MTX).Cyclosporine (CsA):Initiated as a continuous 24-hour intravenous infusion at a dose of 2 mg/kg/day, starting from day -9 before transplantation.Once the patient can tolerate oral intake, cyclosporine is switched to oral administration at a dose of 3-5 mg/kg/day, divided into two daily doses.The target therapeutic trough concentration of cyclosporine should be maintained between 150-250 μg/L.
* Delayed Oral Cyclosporine Protocol:Continue IV infusion until day +20, even if GI symptoms resolve.Switch to oral only if no acute GVHD occurs.If grade II-IV acute GVHD develops, continue IV CsA.

  4.Subsequent Treatment for Patients Unsuitable for or Declining Transplantation 4.1 Consolidation Therapy (Two Cycles)
* Option A Intermediate-Dose Cytarabine-Based Regimen：Liposomal Mitoxantrone: 10 mg/day on days 1-2 (dose-reduced).Cytarabine: 1 g/m² every 12 hours for 3 days (days 1-3).
* Option B VA Regimen (Venetoclax + Azacitidine)：Venetoclax (V): Dose-escalation starting at 100 mg on day 1, increasing to 400 mg/day by day 6, continued through day 14.Azacitidine (A): 75 mg/m²/day subcutaneously or intravenously on days 1-7.
* Treatment Cycle:Each regimen is administered for two cycles with a 3-week interval between cycles, followed by maintenance therapy.

4.2 Maintenance Therapy After Two Consolidation Cycles

* Pegylated Interferon α-2b (Long-acting Interferon): 180μg subcutaneously every two weeks.

Continued until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age: 14 years - 65 years;
* Excluding AML-M3 (Acute Promyelocytic Leukemia) patients;
* Diagnosis conforming to the Chinese Diagnosis and Treatment Guidelines for Adult Acute Myeloid Leukemia (Non-APL) (2023 Edition), including low-risk, intermediate-risk, and high-risk patients;
* Bone marrow morphology indicating hypercellularity or hypocellularity;
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-2.

Exclusion Criteria:

* Presence of intracranial hemorrhage;
* Pregnancy;
* Psychiatric illness or other conditions precluding protocol adherence;
* Severe cardiac arrhythmia, abnormal ECG (QTc >500 ms).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-08-06 (Estimated); Study Completion 2027-08-06 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 24 months
The Complete Response (CR) rate | 24 months
  The Complete Response (CR) rate refers to the proportion of patients achieving complete remission in a treatment regimen.
Partial Response (PR) rate | 24 months
  The Partial Response (PR) rate in oncology indicates the proportion of patients experiencing a significant reduction in tumor size post-treatment.
No Remission (NR) | 24 months
  Non-Response (NR) in medicine refers to the lack of therapeutic response, indicating no significant improvement in a patient's condition post-treatment.
CR with incomplete hematologic recovery (CRi) | 24 months
Therapeutic efficacy | 24 months
  The efficacy of the preparative regimen and anti-GVHD regimen for allogeneic stem cell transplantation in AML patients.

SECONDARY OUTCOMES:
Treatment-Related Mortality (TRM) | 24 months
Overall Survival (OS) | 24 months
Event-Free Survival (EFS) | 24 months
Therapeutic efficacy | 24 months
  The therapeutic efficacy of the integrated protocol, especially for high-risk AML patients (e.g., those harboring FLT3-ITD, IDH1, TP53 mutations, complex karyotype) without the use of targeted agents.
Adverse Event | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China